CLINICAL TRIAL: NCT01973907
Title: Pilot Study for the SQUEEZE Trial: a Trial to Determine Whether Septic Shock Reversal is Quicker in Pediatric Patients Randomized to an Early Goal Directed Fluid-sparing Strategy vs. Usual Care (SQUEEZE)
Brief Title: Pilot Study for the SQUEEZE Trial
Acronym: SQUEEZE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: McMaster Children's Hospital (Other)
Collaborators: Hamilton Health Sciences Corporation (Other); McMaster University (Other); Canadian Critical Care Trials Group (Other)
Responsible Party: Principal Investigator, Melissa J Parker, MD, MSc, Associate Professor of Pediatrics, McMaster University; Staff Physician, McMaster Children's Hospital, McMaster Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13-295
Record Dates: First submitted 2013-10-27; First posted 2013-11-01 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2016-08

CONDITIONS: Septic Shock
Keywords: Sepsis; Septic Shock; Fluid Therapy; Pediatrics; Resuscitation; Emergency Medicine; Critical Care
MeSH Terms: conditions — Shock, Septic; Sepsis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care Resuscitation Strategy (No Intervention): Decisions regarding the IV/IO administration of isotonic fluid boluses and/or the initiation and escalation of vasoactive medication infusions are left to the discretion of the treating physician and medical team. We ask that vasoactive medications not be initiated until at least 60 mL/kg (3 litres for children ≥ 50 kg) of isotonic fluid bolus therapy has been administered. The treating physician and medical team are advised to follow ACCM guidelines for the resuscitation of neonatal and pediatric septic shock and to target ACCM recommended therapeutic endpoints.
- Fluid Sparing Resuscitation Strategy (Experimental): The treating physician and medical team are advised to follow the assigned Fluid Sparing Resuscitation Strategy to guide decisions regarding the IV/IO administration of further isotonic fluid boluses, and the timing of initiation and escalation of vasoactive medication infusions to target the therapeutic endpoints recommended in the ACCM guidelines for the resuscitation of neonatal and pediatric septic shock.
  Interventions: Other: Fluid Sparing Resuscitation Strategy

INTERVENTIONS:
Other: Fluid Sparing Resuscitation Strategy — Tier 1: Initiate IV/IO vasoactive medication infusion support immediately. Further IV/IO isotonic fluid bolus therapy [crystalloid (0.9% Normal Saline or Ringers Lactate) or colloid (5% Albumin)] should be avoided; small volume isotonic fluid boluses [5-10 mL/kg (250-500 mL for participants ≥ 50 kg)] may be provided if required due to A. Clinically unacceptable delay in ability to initiate vasoactive medication infusion(s) and/or 2. Documented intravascular hypovolemia.
  Tier 2: Vasoactive medication(s) should be preferentially titrated/escalated to achieve recommended ACCM hemodynamic goals. Further IV/IO isotonic fluid bolus therapy [crystalloid (0.9% Normal Saline or Ringers Lactate) or colloid (5% Albumin)] should be avoided; small volume isotonic fluid boluses [5-10 mL/kg (250-500 mL for participants ≥ 50 kg)] may be provided if required due to A. Documented intravascular hypovolemia.
  Intervention end: Patient is free from vasoactive medication support and shock is reversed.
  Arms: Fluid Sparing Resuscitation Strategy

SUMMARY:
The purpose of the SQUEEZE Trial is to determine which fluid resuscitation strategy results in the best outcomes for children treated for suspected or confirmed septic shock. In this study, eligible children will be randomized to either the 'Usual Care Arm' or the 'Fluid Sparing Arm'. Children will receive treatment according to current ACCM Septic Shock Resuscitation Guidelines, with the assigned resuscitation strategy used to guide administration of further fluid boluses as well as the timing of initiation and escalation of vasoactive medications to achieve ACCM recommended hemodynamic targets.

DETAILED DESCRIPTION:
Current pediatric surviving sepsis guidelines from the American College of Critical Care Medicine (ACCM) emphasize an early and goal-directed approach to resuscitation. These guidelines suggest that fluid resuscitation should be aggressive with repeated intravenous (IV) fluid boluses of 20 mL/kg, such that some children may require as much as 200 mL/kg of fluid to achieve therapeutic endpoints. The guidelines also recommend the initiation of vasoactive agents at the stage of "fluid refractory shock", i.e. when there is persistent hypoperfusion despite at least 60 ml/kg IV fluid. Improvements in pediatric septic shock survival have been attributed to adherence to the first iteration of the ACCM septic shock guidelines, and the use of goal directed targets. However, the largest and most publicized pediatric trial of fluid resuscitation in children with suspected septic shock (FEAST Trial), published in NEJM in 2011, demonstrated an increased mortality among children treated with aggressive fluid resuscitation in comparison to the conservative fluid resuscitation arm. As a result, the pediatric critical care community clearly acknowledges that these results, while important, are not necessarily generalizable to developed countries such as Canada.

Emerging publications in the ICU literature suggest that excessive compared to conservative fluid administration in adults with septic shock worsens outcomes such as duration of mechanical ventilation, complications related to the third-spacing of fluids, length of ICU stay, and mortality. A systematic review published in August 2012 reveals a paucity of randomized controlled trial (RCT) evidence apart from the FEAST trial examining the impact of fluid resuscitation on mortality in children with septic shock. This raises the important question of whether children in developed countries would also benefit from a fluid sparing resuscitation strategy to achieve the ACCM goal-directed targets. Use of such a fluid sparing strategy would, by default, require earlier initiation and preferential escalation of vasoactive medications to meet ACCM hemodynamic goals. The optimal degree of fluid resuscitation and the timing of initiation of vasoactive support in order to achieve therapeutic targets in children with septic shock remains unanswered.

This Pilot Randomized Controlled Trial constitutes the first step in answering our research question of whether, in pediatric patients with septic shock, use of a fluid sparing strategy to achieve ACCM therapeutic goals, results in improved clinical outcomes without an increased risk of adverse events, compared to the usual care of aggressive fluid resuscitation as currently recommended by the ACCM guidelines. The purpose of the pilot study is to determine feasibility and inform the appropriate methodological design of the larger multi-centre RCT to fully answer our research question. The hypothesis of the pilot study is that the SQUEEZE Trial is feasible to conduct.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for 1 and 3 must be answered YES to be eligible for study.

1. Age 29 days to less than 18 years of age

2a) Patient has Persistent Signs of Shock including one or more of the following: i) Vasoactive Medication Dependence ii) Hypotension (Systolic Blood Pressure and/or Mean Blood Pressure less than the 5th percentile for age) iii) Abnormal Perfusion (2 or more of: abnormal capillary refill, tachycardia, decreased level of consciousness, decreased urine output)

2b) Suspected or Confirmed Septic Shock (Shock due to Suspected or Confirmed Infectious Cause)

2c) Patient has received initial fluid resuscitation of: Minimum of 40 mL/kg of isotonic crystalloid (0.9% Normal Saline and/or Ringer's Lactate) and/or colloid (5% albumin) as fluid boluses within the previous 6 hours for patients weighing less than 50 kg, OR Minimum of 2 litres (2000 mL) of isotonic crystalloid (0.9% Normal Saline and/or Ringer's Lactate) and/or colloid (5% albumin) as fluid boluses within the previous 6 hours for patients weighing 50 kg or more

3. Patient has Fluid Refractory Septic Shock as defined by the Presence of all of 2a, 2b, and 2c.

Exclusion Criteria:

* Patient admitted to the Neonatal Intensive Care Unit (NICU)
* Patient requiring resuscitation in the Operating Room (OR) or Post-Anesthetic Care Unit (PACU)
* Full active resuscitative treatment not within the goals of care
* Shock Secondary to Cause other than Sepsis (i.e. obvious signs of cardiogenic shock, anaphylactic shock, hemorrhagic shock, spinal shock)
* Previous enrolment in this trial, where known by the research team

Ages: 29 Days to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 53 (Actual)
Dates: Start 2014-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Feasibility of conducting the SQUEEZE Trial | The earliest of: 1. Recruitment of the planned 50 participants, or 2. 24 months following initiation of recruitment
  The Primary Outcome of Feasibility of conducting the SQUEEZE Trial will be evaluated based on the following:
  1. Participant enrolment rate: We will define success as an enrolment rate of at least 2 patients/month (recognizing that enrolment may be slower during the study run-in phase).
  2. Protocol adherence: the ability to execute the study procedures. We will assess our ability to initiate study procedures in enrolled patients within 1 hour of randomization.

SECONDARY OUTCOMES:
Appropriateness of eligibility criteria | The earliest of: 1. Recruitment of the planned 50 participants, or 2. 24 months following initiation of recruitment
  We will determine our ability to enroll patients based on the current eligibility criteria, to inform the design of a future multi-centered RCT.
Clinical outcomes | The earliest of: 1. Recruitment of the planned 50 participants, or 2. 24 months following initiation of recruitment
  We will assess our ability to collect clinical outcome data of interest to determine the most appropriate outcomes, perform a sample size calculation, and inform the design of a definitive multi-centered RCT. Clinical outcomes include:
  i) PICU admission rate, PICU Length of Stay, Ventilator Free Days, Acuity Scores (PRISM III), Organ Dysfunction scores (PELOD, PELOD 2), Vasoactive Medication Score, Mortality (28-day, 60-day, and 90-day), Hospital Mortality
  ii) Adverse Events- complications which may be attributable to third spacing of fluid, or inotrope/vasopressor use, including: Intrabdominal Hypertension, Abdominal Compartment Syndrome, Pulmonary Edema, Pleural Effusion requiring drainage, Signs of Digital Ischemia, Digital/Limb Revision amputation, Bowel Ischemia
  iii) Short term hemodynamic outcomes- time to shock reversal determined by freedom from vasoactive medication(s), bedside hemodynamic measurements (HR, MAP, CVP, and non-invasive CO (CI) measurement (USCOM)
Process Feasibility | The earliest of: 1. Recruitment of the planned 50 participants, or 2. 24 months following initiation of recruitment
  We will collect descriptive data related to study Process feasibility to inform conduct of a multi-centred RCT
Resource Feasibility | The earliest of: 1. Recruitment of the planned 50 participants, or 2. 24 months following initiation of recruitment
  We will collect descriptive data related to study Resource feasibility to inform conduct of a multi-centred RCT.
Management Feasibility | The earliest of: 1. Recruitment of the planned 50 participants, or 2. 24 months following initiation of recruitment
  We will collect descriptive data related to study Management feasibility to inform conduct of a multi-centred RCT.

OTHER OUTCOMES:
Daily Fluids | Over the Duration of the Intervention Period, Defined as from the time of Randomization (Time zero) until 24 hours after Shock is Reversed
  We will record daily intake of fluids and blood products and fluid losses to characterize these and calculate daily fluid balance
Fluids Received in the 24 hours prior to study entry | 24 hour period immediately prior to randomization (time zero)
  We will record the intake of fluids and blood products in the 24 hours immediately prior to randomization to characterize these
Positive Culture results from specimens obtained during the Intervention Period | Over the Duration of the Intervention Period, Defined as from the time of Randomization (Time zero) until 24 hours after Shock is Reversed
  We will record daily positive culture results from specimens obtained during the intervention period
Positive Culture Results from specimens obtained in the 24 hours immediately prior to study entry | The 24 hour period immediately prior to Randomization (Time zero)
  We will record positive culture results from specimens obtained in the 24 hours immediately prior to Randomization (Time zero)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa J Parker, MD, MSc, Principal Investigator — McMaster University and McMaster Children's Hospital
Locations (1):
- McMaster Children's Hospital, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
The final trial data set will be made publicly available.

REFERENCES:
- [Derived] Parker MJ, Choong K, Fox-Robichaud A, Liaw PC, Thabane L; Canadian Critical Care Trials Group and the Canadian Critical Care Translational Biology Group. The SQUEEZE pilot trial: a trial to determine whether septic shock reversal is quicker in pediatric patients randomized to an early goal directed fluid-sparing strategy vs. usual care. Pilot Feasibility Stud. 2025 Nov 28;11(1):153. doi: 10.1186/s40814-025-01731-4. PMID 41316443
- [Derived] Parker MJ, Foster G, Fox-Robichaud A, Choong K, Mbuagbaw L, Thabane L; With the SQUEEZE Trial Steering Committee and on behalf of the SQUEEZE Trial Investigators, the Canadian Critical Care Trials Group, Pediatric Emergency Research Canada, and the Canadian Critical Care Translational Biology Group. Statistical analysis plan for the SQUEEZE trial: A trial to determine whether septic shock reversal is quicker in pediatric patients randomized to an early goal-directed fluid-sparing strategy vs. usual care (SQUEEZE). Crit Care Resusc. 2024 Jun 22;26(2):123-134. doi: 10.1016/j.ccrj.2024.02.002. eCollection 2024 Jun. PMID 39072232
- [Derived] Parker MJ, Thabane L, Fox-Robichaud A, Liaw P, Choong K; Canadian Critical Care Trials Group and the Canadian Critical Care Translational Biology Group. A trial to determine whether septic shock-reversal is quicker in pediatric patients randomized to an early goal-directed fluid-sparing strategy versus usual care (SQUEEZE): study protocol for a pilot randomized controlled trial. Trials. 2016 Nov 22;17(1):556. doi: 10.1186/s13063-016-1689-2. PMID 27876084